CLINICAL TRIAL: NCT05854485
Title: Robot-Aided Assessment and Rehabilitation of Upper Extremity Function After Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Kelly Westlake, Associate Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HP-00105650
Record Dates: First submitted 2023-04-18; First posted 2023-05-11 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2024-09

CONDITIONS: Stroke
Keywords: Stroke Rehabilitation; Robotic Rehabilitation; Functional Electrical Stimulation
MeSH Terms: conditions — Stroke | interventions — proto-oncogene protein c-fes-fps; Population Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hybrid multi-muscle FES+Robot (Experimental): Participants will be receive hybrid upper extremity training involving the combination of REACH robotic device and multi-muscle FES. Water based electrodes will be positioned on the Triceps, Anconeus, wrist and finger extensors. Stimulation intensity of FES will be set at the participants tolerance level. The FES induced muscle contraction timing will be triggered in synchrony with the robotic movement. The training will be a multi-directional reach movement and hand opening re-training.
  Interventions: Combination Product: REACH robotic training and multi-muscle Functional Electrical Stimulation (FES) group
- Robot only (Active Comparator): Participants will receive upper extremity training with the REACH robotic device. The training will be a multi-directional reach movement re-training.
  Interventions: Combination Product: Robot only group

INTERVENTIONS:
Combination Product: REACH robotic training and multi-muscle Functional Electrical Stimulation (FES) group — Participants in this group will receive multi-muscle FES during arm robotic training
  Arms: Hybrid multi-muscle FES+Robot
Combination Product: Robot only group — Participants in this group will receive arm robotic training only
  Arms: Robot only

SUMMARY:
The purpose of this clinical trial is to investigate the efficacy of a hybrid-based rehabilitation program for the upper extremity(UE) combining the interventions- Functional Electrical Stimulation (FES) and Robotic rehabilitation in individuals with chronic stroke. The main question it aims to answer is if the Hybrid multi-muscle FES+Robot upper extremity rehabilitation is more effective in improving the upper extremity motor impairments and function as compared to robotic upper extremity training alone.

DETAILED DESCRIPTION:
Individuals with chronic stroke(> 6months after stroke) will be recruited. All participants will complete clinical and kinematic assessments at 2 time points(baseline and after 6 weeks training). Each participant will receive 18 sessions of 60 minute upper extremity training over 6 weeks.

Study participants will be randomly assigned to receive either of the following upper extremity training- 1. Hybrid multi-muscle FES+Robot training group or 2.Robot only training group.

The following clinical assessments to measure the motor impairments and functional recovery will be performed: Fugl-Meyer Upper Extremity, Modified Ashworth Scale, and Wolf Motor Function Test.

Kinematic assessments will be conducted using the REACH robotic device and the Kinereach/trakStar system. The following kinematic parameters will be collected: Smoothness, Range of Motion, and Speed.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals with chronic stroke(>6months post stroke)
2. Age-22-85 years old
3. Ability to perform a Upper Extremity forward reach of about 3 inches

Exclusion Criteria:

1. Upper Extremity co-morbidities-pain, arthritis, and other neurological disorders
2. Unable to tolerate electrical stimulation
3. Have implants such as pacemaker, spinal cord or deep brain stimulator
4. Have an elbow contracture of greater than 150 degrees
5. Receiving Botox injections within 3 months

Ages: 22 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2023-09-06 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Kinematic Assessment:Smoothness in 1/s2 | Change from Baseline Smoothness at 6 weeks
  This measure will be collected as the participants performs target reaching out and in movements of the arm. Smoothness will be collected from the REACH robotic device to determine the kinematic changes in the reaching movements. Kinereach/trakStar system will also be utilized to conduct kinematic assessment and determine the translation of training effects into functional upper extremity use.
Kinematic Assessment:Speed in cm/seconds | Change from Baseline Speed at 6 weeks
  This measure will be collected as the participants performs target reaching out and in movements of the arm. Speed will be collected from the REACH robotic device to determine the kinematic changes in the reaching movements. Kinereach/trakStar system will also be utilized to conduct kinematic assessment and determine the translation of training effects into functional upper extremity use.
Kinematic Assessment:Range of Motion(ROM) in cms | Change from Baseline ROM at 6 weeks
  This measure will be collected as the participants performs target reaching out and in movements of the arm. ROM will be collected from the REACH robotic device to determine the kinematic changes in the reaching movements. Kinereach/trakStar system will also be utilized to conduct kinematic assessment and determine the translation of training effects into functional upper extremity use.

SECONDARY OUTCOMES:
Fugl-Meyer Upper Extremity(FMA-UE) | Change from Baseline FMA-UE at 6 weeks
  FMA-UE is a standard measure for the clinical assessment of motor impairment. FMA mainly evaluates the degree of synergy pattern during volitional movements, along with reflex activity and coordination. It is based on 33 items and scores range from 0 to 66. A higher score means better motor function.
Modified Ashworth Scale of muscle spasticity (MAS) | Change from Baseline MAS at 6 weeks
  The MAS is a measurement of spasticity across specific muscle groups. The grading of spasticity ranges from 0 to 5 with higher score indicating worse functioning.
Wolf Motor Function Test (WMFT) | Change from Baseline WMFT at 6 weeks
  WMFT is a function based test designed to measure upper extremity movements and movement speed during functional tasks. The WMFT consists of 17 items, of which 15 measure time to perform functional tasks and 2 strength-based tasks. Two types of scores are recorded during the task:WMFT-TIME(time of the task) and WMFT-FAS (functional abilities). The maximum score of WMFT-TIME is 120 seconds, and a higher score means slower movement. WMFT-FAS is scored from 0 to 5, and a higher score indicates higher level of functional performance, better quality of the paretic upper extremity during the task.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maryland School of Medicine, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Resquin F, Cuesta Gomez A, Gonzalez-Vargas J, Brunetti F, Torricelli D, Molina Rueda F, Cano de la Cuerda R, Miangolarra JC, Pons JL. Hybrid robotic systems for upper limb rehabilitation after stroke: A review. Med Eng Phys. 2016 Nov;38(11):1279-1288. doi: 10.1016/j.medengphy.2016.09.001. Epub 2016 Sep 29. PMID 27692878
- [Background] Hughes AM, Freeman CT, Burridge JH, Chappell PH, Lewin PL, Rogers E. Feasibility of iterative learning control mediated by functional electrical stimulation for reaching after stroke. Neurorehabil Neural Repair. 2009 Jul-Aug;23(6):559-68. doi: 10.1177/1545968308328718. Epub 2009 Feb 3. PMID 19190087
- [Background] Duret C, Grosmaire AG, Krebs HI. Robot-Assisted Therapy in Upper Extremity Hemiparesis: Overview of an Evidence-Based Approach. Front Neurol. 2019 Apr 24;10:412. doi: 10.3389/fneur.2019.00412. eCollection 2019. PMID 31068898
- [Background] Kahn LE, Zygman ML, Rymer WZ, Reinkensmeyer DJ. Robot-assisted reaching exercise promotes arm movement recovery in chronic hemiparetic stroke: a randomized controlled pilot study. J Neuroeng Rehabil. 2006 Jun 21;3:12. doi: 10.1186/1743-0003-3-12. PMID 16790067
- [Background] Volpe BT, Lynch D, Rykman-Berland A, Ferraro M, Galgano M, Hogan N, Krebs HI. Intensive sensorimotor arm training mediated by therapist or robot improves hemiparesis in patients with chronic stroke. Neurorehabil Neural Repair. 2008 May-Jun;22(3):305-10. doi: 10.1177/1545968307311102. Epub 2008 Jan 9. PMID 18184932
- [Background] Ambrosini E, Zajc J, Ferrante S, Ferrigno G, Gasperina SD, Bulgheroni M, Baccinelli W, Schauer T, Wiesener C, Russold M, Gfoehler M, Puchinger M, Weber M, Becker S, Krakow K, Immick N, Augsten A, Rossini M, Proserpio D, Gasperini G, Molteni F, Pedrocchi A. A Hybrid Robotic System for Arm Training of Stroke Survivors: Concept and First Evaluation. IEEE Trans Biomed Eng. 2019 Dec;66(12):3290-3300. doi: 10.1109/TBME.2019.2900525. Epub 2019 Jun 5. PMID 31180833
- [Background] Collins KC, Kennedy NC, Clark A, Pomeroy VM. Kinematic Components of the Reach-to-Target Movement After Stroke for Focused Rehabilitation Interventions: Systematic Review and Meta-Analysis. Front Neurol. 2018 Jun 25;9:472. doi: 10.3389/fneur.2018.00472. eCollection 2018. PMID 29988530
- [Background] Turner DL, Ramos-Murguialday A, Birbaumer N, Hoffmann U, Luft A. Neurophysiology of robot-mediated training and therapy: a perspective for future use in clinical populations. Front Neurol. 2013 Nov 13;4:184. doi: 10.3389/fneur.2013.00184. PMID 24312073
- [Background] Moon SH, Choi JH, Park SE. The effects of functional electrical stimulation on muscle tone and stiffness of stroke patients. J Phys Ther Sci. 2017 Feb;29(2):238-241. doi: 10.1589/jpts.29.238. Epub 2017 Feb 24. PMID 28265148